CLINICAL TRIAL: NCT05054400
Title: Study of Laser Interstitial Thermal Therapy (LITT) Treatment Response Assessment With Fluciclovine PET MR
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: 0 participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1030
Record Dates: First submitted 2021-09-03; First posted 2021-09-23 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Brain Metastases; Cancer; Gliomas; Glioblastoma
MeSH Terms: conditions — Brain Neoplasms; Neoplasms; Glioma; Glioblastoma | interventions — fluciclovine F-18; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- F18 Fluciclovine (Other): radioactive imaging agent help researchers better "see" how the disease is responding to laser interstitial thermal therapy (LITT)
  Interventions: Drug: F18 Fluciclovine; Other: Standard of Care

INTERVENTIONS:
Drug: F18 Fluciclovine — Given by IV
Other: Standard of Care — Standard of care

SUMMARY:
The purpose of this study is to assess the relationship between brain malignancy volume as defined by post-contrast T1 weighted and F18 Fluciclovine before and following LITT. We hypothesize that imaging with F18 Fluciclovine will be superior to anatomic MR imaging in lesion volume assessment before treatment and that residual F18 Fluciclovine defined tumor will predict local post-LITT disease recurrence.

DETAILED DESCRIPTION:
Primary Objectives

-To estimate the accuracy of F18 Fluciclovine PET MR for laser interstitial thermal therapy (LITT) treatment response assessment as determined by T1 post-contrast MR brain imaging.

Secondary Objectives

* To assess changes in F18 Fluciclovine defined disease with LITT.
* To assess the volume change of the idealized quantitative T1 values of lesions compared -To assess the volume change of idealized quantitative T2 values of lesions compared to -Chemical Exchange Saturation Transfer (CEST) MRI - To assess the ability of CEST imaging to differentiate treatment change from residual disease in brain malignancy following LITT.
* Multiple B Value Diffusion Imaging (Adv Diff) - To assess whether Adv Diff can differentiate treatment changes from residual disease in brain malignancy following LITT.
* Gradient- and Spin-Echo DSC perfusion imaging - To assess whether GESE DSC improves differentiation of treatment change from residual disease in brain malignancy -Adv ASL perfusion imaging - To assess the ability of Adv ASL to differentiate treatment change from residual disease in brain malignancy following radiation therapy.
* Exploratory Objectives
* To assess the relationship between post-LITT enhancing brain tissue and F18 -To assess changes in regional homogeneity (ReHo) values after LITT.

ELIGIBILITY:
Inclusion Criteria

* An adult patient with suspected or pathology-proven central nervous system neoplasm.
* MRI of the brain, positive for at least one intra-axial lesion greater than 5 mm.

Exclusion Criteria

* Contraindication to MR imaging.
* Known allergy to gadolinium-based contrast agents.
* Renal failure as defined by a GFR less than 30 or the use of hemodialysis.
* Pregnant.
* Patients less than 18 years of age will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
To establish the relationship between brain malignancy volume as defined by post-contrast T1 weighted and F18 Fluciclovine before and following LITT. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jason Johnson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org